CLINICAL TRIAL: NCT02514343
Title: Intra-articular Infiltration With Magnesium Sulphate and Bupivacaine in Distal Radius Fractures. Randomized, Double-blind Study
Brief Title: Magnesium Sulfate and Bupivacaine for Rehabilitation After Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Carlos A Acosta-Olivo, MD, PhD, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OR15-009
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Radius Fracture
Keywords: radius fracture; magnesium sulfate; rehabilitation; bupivacaine
MeSH Terms: conditions — Radius Fractures | interventions — Magnesium Sulfate; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium sulfate (Experimental): Will administrate 1 ml of magnesium sulfate 10% and 1.5 mL of sterile water
  Interventions: Drug: Magnesium Sulfate
- Bupivacaine (Experimental): Will administrate 1 ml of magnesium sulfate 10% and 1.5 ml of bupivacaine (5mg/ml)
  Interventions: Drug: Magnesium Sulfate; Drug: Bupivacaine

INTERVENTIONS:
Drug: Magnesium Sulfate — 1ml of 10% magnesium sulfate with 1.5 ml of sterile water
  Other Names: Sulfamag; Epsom Salt
Drug: Bupivacaine — 1.5 ml of Bupivacaine 5mg/ml plus 1 ml of 10% magnesium sulfate
  Other Names: Marcaine; Sensorcaine
  Arms: Bupivacaine

SUMMARY:
This study evaluates the effect of 10% magnesium sulfate in the rehabilitation of the wrist mobility in patients with distal radius fracture treated with percutaneous pinning and plaster

DETAILED DESCRIPTION:
The fractures of distal radius are one of the injuries more frequents in orthopedics. Represent between 8-15% of all bone injuries in adults, and account for up to 20% of all fractures seen in emergency departments.

Despite the frequency of fractures of the distal radius, there is controversy about what is the best way to treat them. The principles of good treatment involving an anatomical reduction with a proper immobilization that keep the reduction. However, the immobilization must be for a brief period to achieve good functional results with a proper rehabilitation, allowing the patient to regain their independence and return to their occupational and daily activities.

One of the treatment employed in the fractures of distal radius is percutaneous pinning and use of rigid immobilization with a plaster for six weeks. Posteriorly we removed the immobilization and percutaneous pins. One of the aspects to take into account is that this procedure is ambulatory and pain in the wrist is an important factor that prevents him from performing a movement joint free, also generating dissatisfaction in the patient.

Recent research has shown that magnesium sulfate reduces postoperative pain applied during the surgical procedure. In addition, it reduces the consumption of opioids and presents no clinical toxicity, for these reasons magnesium sulfate can be considered as an effective adjunct to analgesia postoperative.

The investigators will realize a controlled clinical trial double blind with specific population characteristics, reproducible, prospective, comparative and longitudinal. This study is proposed to study 40 patients, randomly divided into two groups.

Intraarticular infiltration Prior to a detailed explanation of the protocol with signing of the informed consent, be performed intraarticular infiltration with magnesium sulfate alone or in combination with bupivacaine according to the randomization made. The patient will not know the group in which it is assigned, only the doctor who prepare the solution to infiltrate. This procedure will take place after the removal of the immobilization and fixation (plaster and pinning).

With the patient sitting, we realize asepxia with AVAGARD ® for 2 minutes., after this we proceed to intra-articular infiltration of the wrist with sterile technique, will be located by palpation the articular space between structures of the radiocarpal joint. One investigator will infiltrate 1ml of 10% magnesium sulfate with 1.5 ml of sterile water for one group and for the second group will put 1 ml of 10% magnesium sulfate plus 1.5 ml of Bupivacaine 5mg/ml. Posteriorly, another evaluator will perform measurements of range of active motion (ROM) with flexion-extension, radial and ulnar deviation, pronation and supination , as well as grip strength with a hydraulic hand dynamometer (JAMAR ®) and with the visual analog scale (VAS) to assess the pain.

The above mentioned tests shall be the minute one and three after intraarticular infiltration. Then apply PRWE (Patient Rated Wrist Evaluation) and DASH (Disabilities of the Arm, Hand and Shoulder) scales., this scales will apply to two and fourth weeks.

In the sample size calculation, was determined to include 20 patients per group, using a formula of mean differences with a standard deviation of 5 and an expected magnitude of the differences of at least 5 points in the PRWE scale, with a confidence interval of 95, power 80, with a p ˂0. 05 statistically significant β adding the error 20.

ELIGIBILITY:
Inclusion Criteria:

* distal radius fracture treated with percutaneous pinning and plaster
* treated in our institution

Exclusion Criteria:

* allergy to drugs used
* drug use or abuse
* psychiatric disease
* pulmonal, cardiac, pancreatic, renal or hepatic disease
* active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) | At 4 week
  Is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. Developed in 1998 for clinical assessment and is used for specific wrist problems.It is one of the reliable upper extremity outcome instrument

SECONDARY OUTCOMES:
Grip strength | At one minute
  Using a hydraulic dynamometer with the patient with elbow in 90º of flexion and forearm in neutral rotation
Wrist mobility | At 2 weeks
  Mobility in flexion, extension, pronation, supination, cubital and radial deviation using a goniometer
Visual Analogue Scale (VAS) | At minute one
  Measure the maximal pain of the patient
Grip strength | At three minute
  Using a hydraulic dynamometer with the patient with elbow in 90º of flexion and forearm in neutral rotation
Wrist mobility | At 4 week
  Mobility in flexion, extension, pronation, supination, cubital and radial deviation using a goniometer
Visual Analogue Scale | At minute three
  Measurement of the maximal pain of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, MD, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Actually is active this study

REFERENCES:
- [Result] Meena S, Sharma P, Sambharia AK, Dawar A. Fractures of distal radius: an overview. J Family Med Prim Care. 2014 Oct-Dec;3(4):325-32. doi: 10.4103/2249-4863.148101. PMID 25657938
- [Result] Kakar S. Clinical Faceoff: Controversies in the Management of Distal Radius Fractures. Clin Orthop Relat Res. 2015 Oct;473(10):3098-104. doi: 10.1007/s11999-015-4335-5. Epub 2015 May 21. No abstract available. PMID 25995175
- [Result] Gunay C, Oken OF, Yavuz OY, Gunay SH, Atalar H. Which modality is the best choice in distal radius fractures treated with two different Kirschner wire fixation and immobilization techniques? Ulus Travma Acil Cerrahi Derg. 2015 Mar;21(2):119-26. doi: 10.5505/tjtes.2015.55938. PMID 25904273
- [Result] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270
- [Result] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Result] Pereira DF, Natour J, Machado NP, Furtado RN. Effectiveness of intra-articular injection in wrist joints according to triamcinolone hexacetonide dose in rheumatoid arthritis: a randomized controlled double-blind study. Am J Phys Med Rehabil. 2015 Feb;94(2):131-8. doi: 10.1097/PHM.0000000000000174. PMID 25171663